CLINICAL TRIAL: NCT00201409
Title: A Randomized Trial of GM-CSF in Patients With ALI/ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Emory University (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Robert C. Hyzy, MD, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 258; P50HL074024 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will be randomized to receive recombinant human GM-CSF (250 mcg/M2).
  Interventions: Drug: GM-CSF
- 2 (Placebo Comparator): Participants will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo will be administered by slow intravenous infusion once daily for 14 days.
  Arms: 2
Drug: GM-CSF — Recombinant human GM-CSF (250 mcg/M2) will be administered by slow intravenous infusion once daily for 14 days.
  Arms: 1

SUMMARY:
This study will test the hypothesis that administration of granulocyte-macrophage colony stimulating factor (GM-CSF) to patients with acute lung injury/acute respiratory distress syndrome (ALI/ARDS) will improve the clinical course and outcome by shortening the duration of mechanical ventilation for these patients.

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory failure due to ALI/ARDS remains a major health problem, despite significant progress in intensive care unit care and ventilator management. ALI/ARDS is characterized by unacceptably high mortality despite enormous expenditure of health care resources. Survivors face long-term consequences that may affect their quality of life. New therapies are needed to improve early survival and to decrease long-term sequelae of this syndrome. GM-CSF is a naturally occurring cytokine that is present in the normal lung, with important roles in pulmonary homeostasis. GM-CSF is essential for normal maturation and function of alveolar macrophages (resident inflammatory cells that are responsible for initial defense against pneumonia). Alveolar epithelial cells line the gas exchange surface of the lung. Acute lung injury and subsequent abnormal healing is linked to delayed repair of damage to the epithelium following initial injury. This can then lead to pulmonary fibrosis. GM-CSF has potent effects on alveolar epithelial cells, promoting proliferation and limiting epithelial cell death. Thus, GM-CSF has a distinctive combination of activities that make it an excellent candidate for a therapeutic intervention in ALI/ARDS. Preliminary studies for this project demonstrate that GM-CSF can protect experimental animals against acute lung injury, can decrease susceptibility to pneumonia, and is protective against pulmonary fibrosis following acute lung injury. There is extensive experience with the administration of recombinant human GM-CSF to human patients (this biological is approved by the FDA and has been well-tolerated in trials involving critically ill patients). This project is based on the hypothesis that administration of GM-CSF will improve clinical outcomes for patients with ALI/ARDS.

DESIGN NARRATIVE:

With the assent of the attending physician, informed consent will be obtained from the patient or next of kin as soon as possible after case identification. Physiologic measurements and specimen collection will begin at the time of entry into the study. Three days after the patient has met criteria for ALI/ARDS or at entry into the study (whichever is later), he/she will be randomized to receive recombinant human GM-CSF (250 mcg/M2) or placebo, administered by slow intravenous infusion once daily for 14 days.

This study will allow entry of patients who have fulfilled criteria for ALI/ARDS for up to 7 days. Treatment will be initiated after patients have met criteria for at least 3 days. Treatment with GM-CSF may prove both safe and effective within the first 1-2 days of lung injury. However, the present study will not address that question. It is unlikely that the opportunity for improved outcome will be lost by delaying therapy for up to 3 days (based on the proposed mechanisms by which GM-CSF might benefit this patient population). Similarly, the decision to treat for 14 days will allow for improved outcome in patients with non-resolving ARDS by reducing the incidence of ventilator-associated pneumonia and by decreasing pathologic fibroproliferation.

The primary endpoint for this study will be the duration of mechanical ventilation. Additional important endpoints will include changes in the severity of physiologic derangements of respiratory gas exchange, non-respiratory organ failure, and incidence of ventilator-associated pneumonia. Additional assessments designed to determine the mechanism of benefit of GM-CSF treatment will include measures of lung epithelial cell integrity and measures of alveolar macrophage (lung inflammatory cell) function.

ELIGIBILITY:
Inclusion Criteria:

Acute onset of illness with:

* PaO2/FiO2 ratio of less than 300 (ALI) or PaO2/FiO2 ratio of less than 200 (ARDS)
* Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph (infiltrates may be patchy, diffuse, homogeneous, or asymmetric)
* Requirement for positive pressure ventilation via an endotracheal tube
* No clinical evidence of left atrial hypertension (pulmonary arterial wedge pressure measure up to 18 mm Hg)
* First three criteria must occur together within a 24-hour interval

Exclusion criteria:

* Greater than 7 days elapsed following institution of mechanical ventilation
* Pregnancy
* Chronic respiratory failure as defined by any of the following: 1) FEV1 less than 20 ml/kg of PBW; or 2) FEV1/FVC less than 50%
* Chronic hypercapnia or hypoxemia
* Hospitalization within the past 6 months for acute respiratory failure
* Chronic home use of oxygen or mechanical ventilation
* Left ventricular failure as defined by New York Heart Association (NYHA) class IV status
* Neutropenia (absolute neutrophil count less than 1000 cells/mm3)
* History of hematological malignancy or bone marrow transplant
* Entry into other intervention clinical trials
* Decision of the patient or attending physician to forego aggressive care
* Expected survival rate of less than 6 months (based solely on pre-existing medical problems [i.e., poorly controlled neoplasm or other end-stage disease])
* AIDS or known history of HIV infection
* Prednisone (or equivalent) therapy greater than or equal to 20 mg/day for a period of not less than 2 months with treatment continuing within 3 weeks prior to screening
* Cytotoxic therapy within 3 weeks of screening
* Morbid obesity defined as greater than 1 kg/c, body weight
* At risk for increased intracranial pressure that may result from permissive hypercapnia or in whom permissive hypercapnia may be otherwise contraindicated
* Neuromuscular disease that would potentially impact ability to wean from mechanical ventilation
* Receiving extracorporeal membrane oxygenation when meeting screening criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2004-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paine, MD, Study Director — University of Utah and University of Michigan; Robert C. Hyzy, M.D., Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Background] Paine R 3rd, Wilcoxen SE, Morris SB, Sartori C, Baleeiro CE, Matthay MA, Christensen PJ. Transgenic overexpression of granulocyte macrophage-colony stimulating factor in the lung prevents hyperoxic lung injury. Am J Pathol. 2003 Dec;163(6):2397-406. doi: 10.1016/S0002-9440(10)63594-8. PMID 14633611
- [Background] Paine R 3rd, Morris SB, Jin H, Wilcoxen SE, Phare SM, Moore BB, Coffey MJ, Toews GB. Impaired functional activity of alveolar macrophages from GM-CSF-deficient mice. Am J Physiol Lung Cell Mol Physiol. 2001 Nov;281(5):L1210-8. doi: 10.1152/ajplung.2001.281.5.L1210. PMID 11597913
- [Background] Baleeiro CE, Wilcoxen SE, Morris SB, Standiford TJ, Paine R 3rd. Sublethal hyperoxia impairs pulmonary innate immunity. J Immunol. 2003 Jul 15;171(2):955-63. doi: 10.4049/jimmunol.171.2.955. PMID 12847267
- [Background] Presneill JJ, Harris T, Stewart AG, Cade JF, Wilson JW. A randomized phase II trial of granulocyte-macrophage colony-stimulating factor therapy in severe sepsis with respiratory dysfunction. Am J Respir Crit Care Med. 2002 Jul 15;166(2):138-43. doi: 10.1164/rccm.2009005. PMID 12119223
- [Background] Matute-Bello G, Liles WC, Radella F 2nd, Steinberg KP, Ruzinski JT, Hudson LD, Martin TR. Modulation of neutrophil apoptosis by granulocyte colony-stimulating factor and granulocyte/macrophage colony-stimulating factor during the course of acute respiratory distress syndrome. Crit Care Med. 2000 Jan;28(1):1-7. doi: 10.1097/00003246-200001000-00001. PMID 10667491
- [Derived] Spencer-Segal JL, Hyzy RC, Iwashyna TJ, Standiford TJ. Psychiatric Symptoms in Survivors of Acute Respiratory Distress Syndrome. Effects of Age, Sex, and Immune Modulation. Ann Am Thorac Soc. 2017 Jun;14(6):960-967. doi: 10.1513/AnnalsATS.201606-468OC. PMID 28358594
- [Derived] Paine R 3rd, Standiford TJ, Dechert RE, Moss M, Martin GS, Rosenberg AL, Thannickal VJ, Burnham EL, Brown MB, Hyzy RC. A randomized trial of recombinant human granulocyte-macrophage colony stimulating factor for patients with acute lung injury. Crit Care Med. 2012 Jan;40(1):90-7. doi: 10.1097/CCM.0b013e31822d7bf0. PMID 21926600

RESULTS

PARTICIPANT FLOW:
Groups:
- GM-CSF Group: Participants will be randomized to receive recombinant human GM-CSF (250 mcg/M2).
- Placebo Group: Participants will be randomized to receive placebo.
Period: Overall Study
Arm/Group | GM-CSF Group | Placebo Group
Started | 65 | 67
Completed | 64 | 66
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GM-CSF Group | Placebo Group | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (15.6) | 48.3 (13.8) | 48.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 35 | 39 | 74

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days During Days 1-28
Time Frame: Measured at Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GM-CSF Group | Placebo Group
Number analyzed (Participants) | 64 | 66
Days | 10.8 (10.5) | 10.7 (10.3)

2. Secondary Outcome: Oxygenation Index Change at Day 15 From Day 1
Description: The oxygenation index is a calculation used in intensive care medicine to measure the fraction of inspired oxygen (FiO2) and its usage within the body. It is calculated as the fraction of inspired oxygen times Mean airway pressure)/Partial pressure of oxygen in arterial blood Day 15 minus first day drug or placebo administered (Day 1).
Time Frame: Day 1, Day 15
Measure: Mean (Standard Deviation); unit: oxygenation index
Arm/Group | GM-CSF Group | Placebo Group
Number analyzed (Participants) | 64 | 66
oxygenation index | -3.5 (10.4) | -4.6 (4.5)

3. Secondary Outcome: Days Without Organ Failure
Description: Non-respiratory
Time Frame: Measured at Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GM-CSF Group | Placebo Group
Number analyzed (Participants) | 64 | 66
days | 15.7 (11.9) | 12.8 (11.3)

ADVERSE EVENTS:
Arm/Group | GM-CSF Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 31/64 | 34/66
Other Adverse Events (participants affected / at risk) | 39/64 | 39/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Group (N=64) | Placebo Group (N=66)
Sepsis or Multi-organ failure (Immune system disorders) | 11 (11) | 13 (13)
Pulmonary SAE (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 16 (16)
Infection SAE (Infections and infestations) | 7 (7) | 9 (9)
Miscellaneous (General disorders) | 2 (2) | 0 — These events were not documented specifically in the records available
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Group (N=64) | Placebo Group (N=66)
Cardiovascular (Cardiac disorders) | 25 (25) | 25 (25)
Fever (Immune system disorders) | 15 (15) | 11 (11)
GI (Gastrointestinal disorders) | 3 (3) | 5 (5)
Hematologic (Blood and lymphatic system disorders) | 26 (26) | 17 (17)
Infection (Infections and infestations) | 13 (13) | 7 (7)
Neurologic (Nervous system disorders) | 4 (4) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 18 (18)
Renal/Hepatic (Hepatobiliary disorders) | 5 (5) | 8 (8)
Metabolic (Metabolism and nutrition disorders) | 7 (7) | 7 (7)
Miscellaneous (General disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No